CLINICAL TRIAL: NCT04700176
Title: A Multi-Center Phase 2 Study of Daratumumab With Pomalidomide and Dexamethasone in Combination With All-Transretinoic Acid in Patients With Multiple Myeloma Previously Exposed to Daratumumab-Based Regimens
Brief Title: A Study of Daratumumab With Pomalidomide, Dexamethasone, and All-Transretinoic Acid in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020-0280
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; pomalidomide; Tretinoin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) (Experimental): Patients with relapsed or refractory multiple myeloma who have progressed on the combination of Dara + Len + Dex (Cohort A) to be treated with a combination of Dara + Pom + Dex + ATRA (All-Transretinoic Acid)
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: All-trans retinoic acid; Drug: Dexamethasone
- Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B) (Experimental): Patients with relapsed or refractory multiple myeloma who have progressed on the combination of Dara + Pom + Dex (Cohort B) to be treated with a combination of Dara + Pom + Dex + ATRA (All-Transretinoic Acid)
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: All-trans retinoic acid; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — During 28-day treatment cycles, patients will receive Dara 16 mg/kg intravenously (IV) at their current dose upon enrollment onto the study depending on their cycle. They will receive Dara depending on the cycle they are in. If they are on cycles 1-2 then they will receive Dara 16 mg/kg IV on days 1,8,15,22; if they are on cycles 3-6 they will receive Dara 16 mg/kg on days 1 and 15; and if they are on cycle 7 or beyond they will receive Dara 16 mg/kg on day 1.
  Other Names: Darzalex
Drug: Pomalidomide — Pomalidomide will be administered at the patient's currently tolerated dose (4,3, or 2 mg po daily) on days 1-21
  Other Names: Pomalyst
Drug: All-trans retinoic acid — ATRA will be administered in a divided dose of twice daily as an oral formulation at 45mg/m2/day for 3 days. The first administration of ATRA will be given in the morning, two days before the scheduled Dara infusion. The last administration of ATRA will be given in the evening of the day that Dara was administered
  Other Names: ATRA
Drug: Dexamethasone — Dexamethasone will be administered at 40 mg once weekly on days 1,8,15 for patients 75 years old and younger and at 20 mg once weekly on days 1,8,15 for patients older than 75.
  Other Names: Decadron

SUMMARY:
The purpose of this study is to test the safety and efficacy of the study drug daratumumab, when given together with Pomalidomide, Dexamethasone, and All-Transretinoic Acid (ATRA).

DETAILED DESCRIPTION:
This is a multi-institution phase II study of ATRA in combination with fixed dose Daratumumab, Pomalidomide and Dex for a total of 33 patients in patients with relapsed multiple myeloma who have progressed on the combination of Dara + Len + Dex. There will also be an exploratory cohort with an additional 10 patients who have progressed on the combination of Dara + Pom + Dex.

ELIGIBILITY:
Inclusion Criteria:

1. Documented multiple myeloma
2. For cohort A, patients must have been previously exposed to Dara+Len+Dex and must have achieved at least stable disease to this combination.
3. For cohort B, patients must have been exposed to Dara + Pom + Dex and must have achieved at least stable disease to this combination.
4. Histologically confirmed and relapsed multiple myeloma with measurable disease, defined by at least one of the following:

   1. Serum monoclonal protein ≥0.5 g/dL;
   2. Monoclonal protein in the urine on 24-hour electrophoresis ≥200 mg;
   3. Serum immunoglobulin free light chain (FLC) ≥10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal;
   4. New of progressing biopsy proven plasmacytoma on exam or imaging; or
   5. Bone marrow plasma cells ≥20%;
5. Cycle 1 day 1 of study treatment must be within 3 months of last exposure to Daratumumab.
6. Life expectancy >3 months
7. ECOG PS 0-2
8. Age ≥18
9. Adequate organ function, including bone marrow, renal, hepatic, pulmonary, and cardiac function based on the last assessment performed within the Screening Period, defined as:

   1. Absolute neutrophil count (ANC) ≥1,000/μL;
   2. Platelet count ≥50,000/μL, (≥30,000/μL if bone marrow plasma cells are ≥50% of cellularity);
   3. Hemoglobin ≥7.5g/dL;
   4. Creatinine clearance ≥60 mL/min (assessed as glomerular filtration rate using the Cockcroft-Gault formula);
   5. Alanine aminotransferase or aspartate aminotransferase <3 x upper limit of normal (ULN);
   6. Total bilirubin <2 x ULN (except for patients with Gilbert's syndrome confirmed by UGT1A1 mutation);
   7. Left ventricular ejection fraction ≥50% as assessed by echocardiography or multi-gated acquisition (MUGA) scan; and
   8. Must have a minimum level of pulmonary reserve defined as Grade <2 dyspnea and pulse oxygenation ≥92% on room air;
10. Prior to first dose of study drug, a woman must be either:

    * Not of childbearing potential: premenarchal; postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone level >40 IU/L or mIU/mL]); permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
    * Of childbearing potential and practicing a highly effective method of birth control for 4 weeks before initiating study treatment that is consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject) Note: If the childbearing potential changes after start of the study (e.g., woman who is not heterosexually active becomes active, premenarchal woman experiences menarche)
    * a woman must begin a highly effective method of birth control, as described above.
11. A woman of childbearing potential must have 2 negative serum (β human chorionic gonadotropin) or urine pregnancy tests during screening, the first one within 28 days prior to the first dose of study drug and the second within 24 hours prior to the first dose of study drug.
12. A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug.
13. Subjects must be willing and able to adhere to the prohibitions and restrictions specified in this protocol and referenced in the informed consent form (ICF).

Exclusion Criteria:

1. Major concurrent illness or organ dysfunction
2. Active GVHD requiring systemic corticosteroids in a subject who previously received allogeneic-SCT.
3. Cord compression or CNS involvement
4. Recent/Prior active malignancy requiring active therapy 2 years prior to enrollment excluding non-melanoma skin cancer.
5. Prior life-threatening hypersensitivity to daratumumab or an IMiD
6. Plasma cell leukemia
7. Pregnant or lactating females
8. Men donating sperm during study
9. Seropositive for human immunodeficiency virus (HIV)
10. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
11. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
12. Chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) less than 50% of predicted normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noa Biran, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Lee HC. Structure and enzymatic functions of human CD38. Mol Med. 2006 Nov-Dec;12(11-12):317-23. doi: 10.2119/2006-00086.Lee. PMID 17380198
- [Background] Chillemi A, Zaccarello G, Quarona V, Ferracin M, Ghimenti C, Massaia M, Horenstein AL, Malavasi F. Anti-CD38 antibody therapy: windows of opportunity yielded by the functional characteristics of the target molecule. Mol Med. 2013 May 20;19(1):99-108. doi: 10.2119/molmed.2013.00009. PMID 23615966
- [Background] Dimopoulos MA, Oriol A, Nahi H, San-Miguel J, Bahlis NJ, Usmani SZ, Rabin N, Orlowski RZ, Komarnicki M, Suzuki K, Plesner T, Yoon SS, Ben Yehuda D, Richardson PG, Goldschmidt H, Reece D, Lisby S, Khokhar NZ, O'Rourke L, Chiu C, Qin X, Guckert M, Ahmadi T, Moreau P; POLLUX Investigators. Daratumumab, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Oct 6;375(14):1319-1331. doi: 10.1056/NEJMoa1607751. PMID 27705267
- [Background] Chari A, Suvannasankha A, Fay JW, Arnulf B, Kaufman JL, Ifthikharuddin JJ, Weiss BM, Krishnan A, Lentzsch S, Comenzo R, Wang J, Nottage K, Chiu C, Khokhar NZ, Ahmadi T, Lonial S. Daratumumab plus pomalidomide and dexamethasone in relapsed and/or refractory multiple myeloma. Blood. 2017 Aug 24;130(8):974-981. doi: 10.1182/blood-2017-05-785246. Epub 2017 Jun 21. PMID 28637662
- [Background] Nijhof IS, Groen RW, Lokhorst HM, van Kessel B, Bloem AC, van Velzen J, de Jong-Korlaar R, Yuan H, Noort WA, Klein SK, Martens AC, Doshi P, Sasser K, Mutis T, van de Donk NW. Upregulation of CD38 expression on multiple myeloma cells by all-trans retinoic acid improves the efficacy of daratumumab. Leukemia. 2015 Oct;29(10):2039-49. doi: 10.1038/leu.2015.123. Epub 2015 May 15. PMID 25975191
- [Background] Nijhof IS, Casneuf T, van Velzen J, van Kessel B, Axel AE, Syed K, Groen RW, van Duin M, Sonneveld P, Minnema MC, Zweegman S, Chiu C, Bloem AC, Mutis T, Lokhorst HM, Sasser AK, van de Donk NW. CD38 expression and complement inhibitors affect response and resistance to daratumumab therapy in myeloma. Blood. 2016 Aug 18;128(7):959-70. doi: 10.1182/blood-2016-03-703439. Epub 2016 Jun 15. PMID 27307294
- [Background] Dimos JT, Rodolfa KT, Niakan KK, Weisenthal LM, Mitsumoto H, Chung W, Croft GF, Saphier G, Leibel R, Goland R, Wichterle H, Henderson CE, Eggan K. Induced pluripotent stem cells generated from patients with ALS can be differentiated into motor neurons. Science. 2008 Aug 29;321(5893):1218-21. doi: 10.1126/science.1158799. Epub 2008 Jul 31. PMID 18669821
- [Background] Wichterle H, Lieberam I, Porter JA, Jessell TM. Directed differentiation of embryonic stem cells into motor neurons. Cell. 2002 Aug 9;110(3):385-97. doi: 10.1016/s0092-8674(02)00835-8. PMID 12176325
- [Background] Collins SJ. The role of retinoids and retinoic acid receptors in normal hematopoiesis. Leukemia. 2002 Oct;16(10):1896-905. doi: 10.1038/sj.leu.2402718. PMID 12357341
- [Background] Kantarjian HM, Keating MJ, Walters RS, Estey EH, McCredie KB, Smith TL, Dalton WT Jr, Cork A, Trujillo JM, Freireich EJ. Acute promyelocytic leukemia. M.D. Anderson Hospital experience. Am J Med. 1986 May;80(5):789-97. doi: 10.1016/0002-9343(86)90617-0. PMID 3458366
- [Background] Cordonnier C, Vernant JP, Brun B, Heilmann MG, Kuentz M, Bierling P, Farcet JP, Rodet M, Duedari N, Imbert M, et al. Acute promyelocytic leukemia in 57 previously untreated patients. Cancer. 1985 Jan 1;55(1):18-25. doi: 10.1002/1097-0142(19850101)55:13.0.co;2-b. PMID 3855265
- [Background] Tallman MS, Kwaan HC. Reassessing the hemostatic disorder associated with acute promyelocytic leukemia. Blood. 1992 Feb 1;79(3):543-53. No abstract available. PMID 1732003
- [Background] Chomienne C, Ballerini P, Balitrand N, Daniel MT, Fenaux P, Castaigne S, Degos L. All-trans retinoic acid in acute promyelocytic leukemias. II. In vitro studies: structure-function relationship. Blood. 1990 Nov 1;76(9):1710-7. PMID 2224120
- [Background] Tallman MS, Andersen JW, Schiffer CA, Appelbaum FR, Feusner JH, Ogden A, Shepherd L, Willman C, Bloomfield CD, Rowe JM, Wiernik PH. All-trans-retinoic acid in acute promyelocytic leukemia. N Engl J Med. 1997 Oct 9;337(15):1021-8. doi: 10.1056/NEJM199710093371501. PMID 9321529
- [Background] Ogata A, Nishimoto N, Shima Y, Yoshizaki K, Kishimoto T. Inhibitory effect of all-trans retinoic acid on the growth of freshly isolated myeloma cells via interference with interleukin-6 signal transduction. Blood. 1994 Nov 1;84(9):3040-6. PMID 7949175
- [Background] Siegel D, Niesvizky R, Miller WH Jr, Busquets X, Kumar R, MIchaeli J: All trans retinoic acid (ATRA) and interferon alfa (IFNa) synergistically inhibit myeloma cell growth and induce retinoic acid receptor alfa (RARa) expression. Blood 80:121a:1992 (abstr, supple 1).
- [Background] Musto P, Falcone A, Sajeva MR, D'Arena G, Bonini A, Carotenuto M. All-trans retinoic acid for advanced multiple myeloma. Blood. 1995 Jun 15;85(12):3769-70. No abstract available. PMID 7780162
- [Background] Frerichs KA et al, Efficacy and safety of daratumumab combined with all-trans retinoic acid in relapsed/refractory multiple myeloma: results of the Phase ½ Dara/Atra study. Blood (2019) 134 S:1:1826.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients enrolled in Cohort B
Groups:
- Total: Total of all reporting groups
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Cohort A)
Description: To determine the ORR of the combination of Dara + Pom + Dex + ATRA in patients progressing on Dara + Len + Dex (Cohort A)
Time Frame: 12 Months
Population: No patients enrolled in Cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

2. Primary Outcome: Incidence of Adverse Events
Description: Incidence of Adverse Events in the combination of Dara + Pom + Dex + ATRA using CTCAE V5 criteria.
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

3. Secondary Outcome: Objective Response Rate (Cohort B)
Description: To determine the ORR of the combination of Dara + Pom + Dex + ATRA in patients progressing on Dara + Pom + Dex
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Arm/Group | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Stringent Complete Response
Description: To determine the best stringent complete response (sCR)/CR/near CR (nCR) and >/= very good partial response (VGPR) rates.
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

5. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: To define the toxicity using CTCAE V5 criteria.
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

6. Secondary Outcome: Rate of Minimal Residual Disease Evaluation
Description: To evaluate the status of minimal residual disease (MRD) in patients who achieve sCR, CR, or nCR.
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

7. Secondary Outcome: Time on Study (TOS)
Description: Duration from start of study treatment to end of study
Time Frame: 12 Months
Population: Patient withdrew consent to follow up at time of progression. No participants enrolled in cohort B
Measure: Number; unit: Months
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Months | 8 |

8. Secondary Outcome: Duration of Response (DOR)
Description: Duration from treatment response to progression
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Measure: Number; unit: Months
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Months | 8 |

9. Secondary Outcome: Time To Progression (TTP)
Description: Duration from start of study treatment to progression
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Measure: Number; unit: Months
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Months | 8 |

10. Secondary Outcome: Progression-Free Survival (PFS)
Description: Duration from start of study treatment to PD or death [regardless of cause], whichever comes first
Time Frame: 12 Months
Population: No participants enrolled in cohort B
Measure: Number; unit: Months
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 1 | 0
Months | 8 |

11. Secondary Outcome: Overall Survival (OS)
Description: Duration from start of study treatment to death
Time Frame: 12 Months
Population: Patient withdrew consent to follow up at time of progression
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are captured from time of consent through 30 days after the last dose of study drug, approximately 8 months
Description: Cohort B was not enrolled
Arm/Group | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) (N=1) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B) (N=0)
Fever (Investigations) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
RSV (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progressed on Daratumumab + Lenalidomide + Dexamethasone (Cohort A) (N=1) | Progressed on Daratumumab + Pomalidomide + Dexamethasone (Cohort B) (N=0)
Brain Fogginess (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation Intermittent (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (7) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RSV (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT04700176/Prot_SAP_000.pdf